CLINICAL TRIAL: NCT00263029
Title: Pre-operative Radiotherapy/ Oxaliplatin/ Capecitabine Treatment For Unresectable Locally-advanced Rectal Cancer (PROCTFUL)
Brief Title: Preoperative Radiotherapy/ Oxaliplatin/ Capecitabine Treatment For Unresectable Locally-advanced Rectal Cancer
Acronym: PROCTFUL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8479
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Oxaliplatin — 60mg/m² as a 2-hour intravenous infusion every week for 5-6 week
Drug: Capecitabine — 500mg tablets and 150mg tablets. 750mg/m² bd given approximately 12 hours apart
Radiation: Radiotherapy — Planned total dose of 45-50.4Gy (with cone down) in 25-28 fractions

SUMMARY:
The purpose of this phase II trial is to determine the efficacy and safety of the combination of oxaliplatin, capecitabine and radiotherapy as preoperative therapy in locally advanced cancers of the rectum.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status score 0-1.
* Chemo-naïve patients.
* Histologically/cytologically confirmed diagnosis of rectal adenocarcinoma (clinically stage mT3 or mT4), either considered (1)inoperable, or (2)locally advanced, where histologically confirmed curative resection is considered unlikely.
* Evaluable measurable disease on imaging with MRI/CT to allow for response assessment.
* Adequate haematological, renal and liver functions as follows:

  * ANC > 3000ml
  * Platelet count > 100,000 ml
  * Urea & Serum Creatinine < 1.5 X upper limit of normal value
  * Total serum bilirubin < 1.5 X upper limit of normal value
  * ALT & AST < 3 X upper limit of normal value

Exclusion Criteria:

* Prior chemotherapy.
* Documented allergy to oxaliplatin or capecitabine.
* Prior radiotherapy to pelvis.
* Previous or concurrent malignancies at other sites with the exception of basal or squamous cell carcinoma of the skin.
* Pregnant or lactating females (with negative pregnancy test documentation in pre-menopausal female patients).
* Currently participating into another clinical trial with any investigational drug in the previous 30 days.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-06; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Response rate (both clinical and pathological) of the primary rectal cancer observed after the chemoradiotherapy. Histologically confirmed complete resection rate (R0 rate). | 3-years disease- free-survival or 3-years overall survival

SECONDARY OUTCOMES:
Adverse events collection | From the signature of the informed consent up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Iris CHAN, MD, Study Director — Sanofi